CLINICAL TRIAL: NCT05662579
Title: Effect of a Core Muscle Resistance Program on Great Trochanteric Pain Syndrome (GTPS): Randomized Clinical Trial
Brief Title: Core Resistance and Lateral Hip Pain
Acronym: GTPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Resistência do core no quadril
Record Dates: First submitted 2022-03-07; First posted 2022-12-22 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Trochanteric Bursitis
Keywords: lateral hip pain; trochanteric bursitis; gluteus medius tendinosis; greater trochanteric gluteal syndrome
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomized blind clinical trial, with a longitudinal characteristic in the area of physiotherapy, orthopedics, postural control and biomechanics. The intervention will consist of 4 weeks, 2 times a week, and the variables of interest will be measured in the pre-treatment period, after 4 weeks (immediately after the end of the protocol) and in the follow up of 12 weeks after the end of the protocol.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluations of the participants and the analysis of the data will be carried out by a researcher blind to the allocation of the subjects in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hip exercises (Experimental): PHASE I: (sessions 1 to 4)
  1. Active exercise without weight support (standing) for abductors, adductors, hip flexors and extensors
  2. Hip extension exercise in 4 supports
  3. Hip abduction exercise in 4 supports ("hydrant")
  4. Oyster Exercise
  5. Hip abduction exercise in lateral decubitus
  6. Hip extension exercise in ventral decubitus
  PHASE II: (sessions 5 to 8)
  1. Hip abduction exercise in lateral decubitus
  2. Progressive resistance exercise for abductors, adductors, flexors and hip extensors with standing theraband
  3. Side walk with theraband positioned at the ankle joint
  4. Squat exercise
  5. Advance exercise
  6. Step down exercise
  Interventions: Other: Exercises
- hip + core exercises (Experimental): In addition to all the exercises in the "hip exercise" group, this group will do:
  PHASE I: (sessions 1 to 4)
  1. Exercise for contraction of the transversus abdominais in the supine position
  2. Bridge exercise
  3. Plank exercise PHASE II: (sessions 5 to 8)
  1. Unilateral bridge exercise 2. Plank exercise with hip extension 3. Lateral plank exercise
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — There will be 2 reevaluations of the participants, similar to the initial: at the end of the exercise protocol and in a follow-up of 12 weeks after the end of the protocol.
  The contraction phase of each exercise will be 2 concentric seconds, 1 isometric second and 2 eccentric seconds, followed by 1 second of rest; there will be approximately 90 seconds of rest between each set of 10 repetitions, time the other member will be exercising.
  At the beginning and at the end of each session, the participants will be asked to point out the pain they feel in the hip at that time. In each of the 8 sessions, the physiotherapist will take note of the presence, lateral pain in the hip at the beginning and end of the therapy (by VAS), number of repetitions performed in each exercise (for the group that will do core exercises, it will be noted the time in seconds of each exercise) and any adverse events. Each series of exercises will be repeated 3 times, all performed bilaterally.

SUMMARY:
Although the middle gluteal muscle is an important stabilizer of the pelvis, no relationship has yet been described between the Great Trochanteric Pain Syndrome (GTPS) and the resistance of the core muscles. Objective: To evaluate the effect of a core resistance program on pain, activation and muscle strength, quality of life and postural control in women with GTPS. Materials and methods: The sample will consist of 36 postmenopausal women with clinical diagnosis of GTPS, who will be randomized into 2 groups: group 1 (hip exercises) and group 2 (hip + core exercises). The treatment protocol will be performed twice a week, for 4 weeks. The same evaluation will be done in 3 moments (in the pre-treatment period, after 4 weeks and 12 weeks after the end of treatment, as a follow up), and will consist of the following analyzes: quality of life (Hip Outcome Score - HOS questionnaire), GTPS severity (VISA-G questionnaire), muscle activation (electromyography - EMG), dynamic postural control (force platform - CoP), muscle strength (load cell), core resistance (supine bridge test and prone bridge test) and pain intensity (Visual Analogue Scale). Expected results: It is intended to establish the effect of a resistance program of core muscles on pain, activation and muscle strength, quality of life and postural control in women with SDGT.

DETAILED DESCRIPTION:
If a patient is using an anti-inflammatory, guided by the orthopedist, or a physiotherapy treatment protocol, start only 10 days after the end of the same. As participants, they will be instructed to avoid activities that cause pain during the research period. All others selected until the final evaluation will be discouraged. For all groups, the use of analytical medication prescribed by the orthopedist will be allowed, when requested. As the participants will be asked each session about the use of their analog, the data and the dosage that will occur during the study period will be noted. If necessary, how researchers will contact the orthopedist for information and guidance. If a participant needs to use anti-inflammatory medication during a survey, they will be excluded.

The analyzes will be carried out by a blind researcher regarding the allocation of the subjects in each group. Participants who have missing data and those who do not attend all treatment sessions will be included in the analysis.

To establish the results, the following variables will be considered:

* Pain intensity: VAS
* Quality of life: scores on the HOS questionnaire
* Severity of symptoms: VISA-G questionnaire
* Muscle activation: (peak of RMS) of the gluteus medius, gluteus maximus, spine erector, rectus abdominis, external oblique, internal oblique / transverse abdominal muscles
* Postural control: elliptical area of the center of pressure oscillation (COP), amplitude of oscillation of the COP and oscillation speed of the COP
* Muscle strength: measurements carried out by the load cell for the abductor, adductor, internal and external rotator groups, extensors, and hip flexors (in Kgf)
* Time (in months) reporting pain in the hip (sample characterization questionnaire)
* Presence or not of hip pain when lying in DL on it (questionnaire to characterize the sample)
* Hours of weekly physical activity (sample characterization questionnaire)
* Use or not of hormone replacement (sample characterization questionnaire)

The Shapiro-Wilk test will be applied to determine the normality of the sample. Student's t test will be used to compare age, weight, height, body mass index (BMI), duration of current illness, level of physical activity, use of hormone replacement and the presence of pain when lying on the hip between groups. The two-way ANOVA test (with Bonferroni post-test) will be used to compare the intra-group and intergroup results, if the data are normal, and will be described as mean and standard deviation. Cohen's D test will be performed to calculate the effect size. Linear correlation between variables will be investigated by Pearson's (or Spearman's) correlation test. If there is a linear correlation between any of the potentially confounding variables, analysis of covariance will be performed using the ANCOVA test. Other necessary analyzes may still be included. The level of statistical significance will be set at p ≤ 0.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal status (amenorrhea for at least 12 months or hysterectomy)
* lateral pain in the hip for at least 3 months
* clinical diagnosis of GTPS performed by an orthopedist

Exclusion Criteria:

* surgery on lower limbs or spine in the last 12 months
* symptoms of osteoarthritis or intra-articular disease of the hip (joint block, limited range of motion and difficulty handling socks and clothes)
* infiltration of the hip with corticosteroids in the last 6 months
* have received physical therapy for this condition in the past 12 months
* participants who need to use anti-inflammatory drugs

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
initial postural control | before starting treatment
  The center of pressure oscillation will be evaluated (COP). The results will be presented in cm2.
Postural control after treatment | immediately after the end of treatment
  The center of pressure oscillation will be evaluated (COP). The results will be presented in cm2.
Postural control after 12 weeks | 12 weeks after the end of treatment
  The center of pressure oscillation will be evaluated (COP). The results will be presented in cm2.
initial Muscle Ativation | before starting treatment
  Muscle activation will be evaluated by surface electromyography and presented in RMS.
Muscle Ativation after treatment | immediately after the end of treatment
  Muscle activation will be evaluated by surface electromyography and presented in RMS.
Muscle Ativation after 12 weeks | 12 weeks after the end of treatment
  Muscle activation will be evaluated by surface electromyography and presented in RMS.

SECONDARY OUTCOMES:
change in hip function | evaluation before treatment, immediately at the end of treatment and after 12 weeks
  In each assessment, participants will respond to the Hip Outcome Score (HOS). The Hip Outcome Score (HOS) is an instrument capable of evaluating physically active patients with hip diseases, without severe degenerative changes. Higher scores mean better functionality. The HOS is a self-administered questionnaire, which has 28 items (questions) divided into two subscales, one for Activities of Daily Living (ADL), with 19 items; and another for Sport, with nine items. Each subscale can vary the final score (score) between 0 and 100, with higher scores representing better hip function.
change in severity of Symptoms | evaluation before treatment, immediately at the end of treatment and after 12 weeks
  at each assessment, participants will respond to the VISA tendinopathy questionnaire for greater trochanteric pain syndrome, the VISA-G. It consists of eight questions that assess current symptoms with total scores ranging from 0 to 100, with higher scores indicating less pain and better function.
change in Core Strenght | evaluation before treatment, immediately at the end of treatment and after 12 weeks
  The time spent in the Prone Bridge Test (in the prone position) will be evaluated in seconds.
change in Muscle Strenght | evaluation before treatment, immediately at the end of treatment and after 12 weeks
  The muscular strength of abductor groups, adductors, internal rotators, hip flexors and extensors will be quantified in kilograms, accessed by load cell. The results will be presented in kilograms.
change in pain intensity | evaluation before treatment, immediately at the end of treatment and after 12 weeks
  the intensity of your pain using the Visual Analog Pain Scale (VAS), which scores your current pain with scores between 0 and 10. Zero is no pain and 10 is considered unbearable pain

CONTACTS AND LOCATIONS:
Locations (1):
- State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Ekstrom RA, Donatelli RA, Carp KC. Electromyographic analysis of core trunk, hip, and thigh muscles during 9 rehabilitation exercises. J Orthop Sports Phys Ther. 2007 Dec;37(12):754-62. doi: 10.2519/jospt.2007.2471. Epub 2007 Aug 29. PMID 18560185
- [Background] Fearon AM, Scarvell JM, Neeman T, Cook JL, Cormick W, Smith PN. Greater trochanteric pain syndrome: defining the clinical syndrome. Br J Sports Med. 2013 Jul;47(10):649-53. doi: 10.1136/bjsports-2012-091565. Epub 2012 Sep 14. PMID 22983121
- [Background] Marshall PW, Murphy BA. Core stability exercises on and off a Swiss ball. Arch Phys Med Rehabil. 2005 Feb;86(2):242-9. doi: 10.1016/j.apmr.2004.05.004. PMID 15706550
- [Background] Ganderton C, Semciw A, Cook J, Pizzari T. Demystifying the Clinical Diagnosis of Greater Trochanteric Pain Syndrome in Women. J Womens Health (Larchmt). 2017 Jun;26(6):633-643. doi: 10.1089/jwh.2016.5889. Epub 2017 Mar 6. PMID 28263673
- [Background] Mallow M, Nazarian LN. Greater trochanteric pain syndrome diagnosis and treatment. Phys Med Rehabil Clin N Am. 2014 May;25(2):279-89. doi: 10.1016/j.pmr.2014.01.009. Epub 2014 Mar 18. PMID 24787333
- [Background] Reid D. The management of greater trochanteric pain syndrome: A systematic literature review. J Orthop. 2016 Jan 22;13(1):15-28. doi: 10.1016/j.jor.2015.12.006. eCollection 2016 Mar. PMID 26955229
- [Background] Del Buono A, Papalia R, Khanduja V, Denaro V, Maffulli N. Management of the greater trochanteric pain syndrome: a systematic review. Br Med Bull. 2012 Jun;102:115-31. doi: 10.1093/bmb/ldr038. Epub 2011 Sep 4. PMID 21893483
- [Background] Rompe JD, Segal NA, Cacchio A, Furia JP, Morral A, Maffulli N. Home training, local corticosteroid injection, or radial shock wave therapy for greater trochanter pain syndrome. Am J Sports Med. 2009 Oct;37(10):1981-90. doi: 10.1177/0363546509334374. Epub 2009 May 13. PMID 19439758